CLINICAL TRIAL: NCT04112797
Title: Prospective Observational Study to Evaluate the Safety of Treatment With A"LLERGOVAC® HIMENÓPTEROS" in Patients Sensitized to This Venom
Brief Title: Study to Evaluate the Safety of Treatment With A"LLERGOVAC® HIMENÓPTEROS" in Patients Sensitized to This Venom
Acronym: HIPNOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: ROX-ALE-2018-02
Record Dates: First submitted 2019-06-18; First posted 2019-10-02 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Allergy to Himenoptera Venom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Allergovac himenoptera — Treatment with allergy vaccine againts Apis mellifera, Vespula spp or Polistes dominula

SUMMARY:
It is a safety and tolerability study of Allergovac Himenopteros in patients sensitized to Apis mellifera, Polistes Dominula or Vespula spp. To get this aim all adverse reactions will be recorded through the study. In addition, it will be evaluated the treatment efficacy with the re-sting after a year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients over 14 years of age with allergy to bee venom, Polistes or Vespula. To meet this criteria, patients must present a systemic reaction with the bite of one of these insects, plus specific IgE detection in the skin test and / or IgE against the himenoptera venom.

  2. Prescription treatment with Hymenoptera venom must be indicated and patients are susceptible to receive Allergovac® Hymenoptera, according to usual clinical practice.

  3. Patients who have given their written consent. In the case of minors, the assent will always be signed by the parent / legal guardian, in addition to the minor.

Exclusion Criteria:

1. Patients who have received treatment with Allergovac® Hymenoptera prior to inclusion in the study.
2. Patients under treatment with immunotherapy against aeroallergens.
3. Patients who have received previous treatment with immunotherapy, with any of the venoms that they are going to receive, in the 5 years prior to the inclusion in the study.
4. Patients who under investigator opinion may present difficulties that prevent the comprehension of what was written in the information sheet for the patient, the informed consent or the completion of self-administered questionnaires.
5. Patients who are participating in another clinical trial or observational study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with allergy to himenoptera venom.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by WAO classification | During 1 year
  All adverse events ocurred during the study Will be collected and clasified following the WAO recommendations. The percentages Will be exposed by number of patients and by dose administrations.

SECONDARY OUTCOMES:
Efficacy of vaccine evaluating re-sting test | Result of the re-sting test
  Grade of treatment protection after controlled sting

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Vega Baja Orihuela, Orihuela, Alicante
  - Hospital Mexoeiro, Vigo, Pontevedra
  - C.H.U. A Coruña, A Coruña
  - Hospital Santa Maria, Lleida
  - Hospital Fundación Alcorcón, Madrid
  - Hospital Universitario Reina Sofia, Murcia
  - Hospital Joan XXIII, Tarragona
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided